CLINICAL TRIAL: NCT00748592
Title: PD 0200390 Dose-Ranging Trial: A Randomized, Double-Blind, Placebo-Controlled, 4-Way Crossover, Multicenter Polysomnography Trial Of PD 0200390 In Elderly Subjects With Primary Insomnia
Brief Title: A Dose-Ranging, Multicenter Polysomnography Trial of PD 0200390 in Elderly Subjects With Primary Insomnia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A4251026
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Insomnia
Keywords: Insomnia, Primary Insomnia, Chronic Insomnia, DIMS (Disorders of Initiating and Maintaining Sleep), Disorders of Initiating and Maintaining Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — (1-aminomethyl-3,4-dimethylcyclopentyl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PD 0200390, 5 mg (Experimental)
  Interventions: Drug: PD 0200390
- PD 0200390, 15 mg (Experimental)
  Interventions: Drug: PD 0200390
- PD 0200390, 30 mg (Experimental)
  Interventions: Drug: PD 0200390

INTERVENTIONS:
Drug: Placebo — Subjects in this arm will be administered 3 capsules of placebo 30 minutes before bedtime for two consecutive nights in the sleep lab.
  Arms: Placebo
Drug: PD 0200390 — Subjects in this arm will be administered 3 capsules totaling 5 milligrams 30 minutes before bedtime for two consecutive nights in the sleep lab.
  Arms: PD 0200390, 5 mg
Drug: PD 0200390 — Subjects in this arm will be administered 3 capsules totaling 15 milligrams 30 minutes before bedtime for two consecutive nights in the sleep lab.
  Arms: PD 0200390, 15 mg
Drug: PD 0200390 — Subjects in this arm will be administered 3 capsules totaling 30 milligrams 30 minutes before bedtime for two consecutive nights in the sleep lab.
  Arms: PD 0200390, 30 mg

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter trial with a 4-way crossover design. Elderly subjects with primary insomnia who meet screening requirements will initially be randomized into the study and receive the first of 4 treatments (PD 0200390 5 mg, 15 mg and 30 mg or placebo) daily 30 minutes before bed time for 2 consecutive days in a polysomnography (PSG) lab.

ELIGIBILITY:
Inclusion Criteria:

* 3 month history of primary insomnia
* Difficulty initiating and maintaining sleep for at least 3 nights/week for the past month (difficulty falling asleep, difficulty staying asleep, early awakening)

Exclusion Criteria:

* Any history of psychiatric diagnosis
* History or presence of any breathing related sleep disorder
* History or presence of any medical or neurological condition that could interfere with sleep
* Use of alcohol as a sleep aid or more than 2 standard drinks consumed per day or more than 14 consumed per week

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Wake After Sleep Onset (WASO) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23

SECONDARY OUTCOMES:
Sleep and early morning behavior as determined by Leeds Sleep Evaluation Questionnaire (LSEQ) | Days -6, -5, 2, 3, 9, 10, 16, 17, 23, and 24
Latency to persistent sleep (LPS) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Latency to REM Sleep as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Sleep efficiency (SE) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Number of awakenings after sleep onset (NAASO) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Total wake time (TWT) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Next day sleepiness as determined by Visual Analog Scale (VAS) for Sleepiness | Days -6, -5, 2, 3, 9, 10, 16, 17, 23, and 24
Number of arousals as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Total sleep time (TST) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Next day performance sa determined by Digit Symbol Substitution Test (DSST) | Days -6, -5, 2, 3, 9, 10, 16, 17, 23, and 24
Subjective Sleep Onset and Maintenance as determined by Subjective Sleep Questionnaire (SSQ) | Days -6, -5, 2, 3, 9, 10, 16, 17, 23, and 24
Wake time during sleep (WTDS) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Wake time after sleep (WTAS) as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Percentages of Stage 1 Sleep, Stage 2 Sleep, Stage 3+4 Sleep, Stage REM Sleep as determined by PSG assessment | Days -7, -6, 1, 2, 8, 9, 15, 16, 22, and 23
Restorative sleep as determined by Restorative Sleep Questionnaire Daily (RSQ D) | Days -6, -5, 2, 3, 9, 10, 16, 17, 23, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4251026&StudyName=A%20Dose-Ranging%2C%20Multicenter%20Polysomnography%20Trial%20of%20PD%200200390%20in%20Elderly%20Subjects%20With%20Primary%20Insomnia%0A